CLINICAL TRIAL: NCT04207528
Title: The Effects of Prosocial Writing on Psychological Well-being: A Randomized Controlled Trial Among Young Adults
Brief Title: Campus Life Study: Harnessing Generativity Among Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Marcie D. Haydon, MA, CPhil, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB#19-002092
Record Dates: First submitted 2019-12-13; First posted 2019-12-23 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Healthy Young Adults
MeSH Terms: interventions — Functional Laterality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Helping Condition (Experimental): Participants in the peer helping condition will be asked to write about their experiences in their first-year at UCLA (freshman or first-year after post-transfer), with an emphasis on using the experience to benefit someone who is about to be a first-year student.
  Interventions: Behavioral: Writing
- Facts-only Control (Active Comparator): Participants in the facts-only writing condition will be asked to write facts about their experiences in their first-year at UCLA (freshman or first-year post-transfer). Unlike the previous conditions, they will not be instructed to write for the benefit of another individual.
  Interventions: Behavioral: Writing

INTERVENTIONS:
Behavioral: Writing — After completing the baseline questionnaire, participants will be randomized to one of two conditions-a peer helping condition or a facts-only writing control. Participants will receive general instructions for completing the writing sessions and will be asked to write for at least 5 minutes per session. Topics covered in each session will vary and are related to common themes relating to life as a first-year university student (e.g., academics, adjusting to university, etc.). Participants will be instructed not to worry about grammar, spelling, or sentence structure and reminded that their responses will remain anonymous. Writing sessions (four in total) will be spaced 1 day apart and take place all within the same week.

SUMMARY:
Recent research suggests that short, online interventions can enhance well-being, which is beneficial to both physical and mental health outcomes. Further, growing evidence suggests that prosocial behavior-a behavior that can be reliably manipulated through a short online intervention-may have beneficial effects on well-being and physical health. Giving support to others appears to be just as beneficial as receiving support, and asking people to perform kind acts for others over the course of several weeks, for example, has been shown to both increase well-being and reduce the inflammatory potential of immune cells.

The purpose of the current study is to test a novel 3-week, online prosocial writing-based intervention in a sample of young adults. Previous intervention studies have manipulated prosocial behavior by asking participants to perform tangible acts of kindness for others, such as writing a note to a coworker or helping a neighbor. However, providing this type of direct support can be logistically challenging and may contribute to increased feelings of distress in certain contexts. Writing interventions designed to elicit feelings of generativity offer one alternative approach, though they have yet to be tested among young adults.

Participants (n = 200) will be randomized to one of two conditions--peer helping or a facts-only control--and instructed to write about their experiences in their first-year at UCLA (freshman or first-year after transfer). Those in the peer helping will be asked to write for the benefit of a student who is about to begin their first year, whereas those in the facts-only control will not. In total, participants will complete 4 writing assignments, each on a separate day over the course of one week. Valid self-report measures will be assessed at pre-intervention, each writing session, post-intervention, and at the 2-week follow-up. The investigators expect participants in the peer helping condition to experience a greater increase in well-being (primary outcome) across the intervention and the follow-up when compared to the control condition. Secondary outcomes will include depressive symptoms, anxiety, loneliness, physical symptoms, social support, and generativity. As an exploratory aim, will also assess several moderators (i.e., psychological distress, prosocial tendencies, generativity) and mediators (i.e., fulfillment of psychological needs, positive affect) of the intervention effects.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in an upper-division psychology course
* 18 years of age or older
* fluent in English
* access to the internet and email

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Change in psychological well-being | At the baseline survey (1 day before the intervention begins), at the post-intervention survey (2 days after the final writing assignment), and and at the 2-week follow-up
  Well-being within the past week will be measured at baseline, post-intervention, and the 2-week follow-up via the 14-item Mental Health Continuum-Short Form (MHC-SF). The MHC-SF is comprised of three empirically derived subscales: the 3-item Emotional Well-Being Subscale, the 6-item Psychological Well-Being Subscale, and the 5-item Social Well-Being Subscale. Higher scores on each subscale, and the total score overall (range: 0-56), indicate greater well-being.

SECONDARY OUTCOMES:
Change in depressive symptoms | At the baseline survey (1 day before the intervention begins), at the post-intervention survey (2 days after the final writing assignment), and and at the 2-week follow-up
  Depressive symptoms over the past week will be measured at baseline, post-intervention, and the 2-week follow-up via the 20-item Center for Epidemiological Studies Depression Scale (CES-D). The CES-D is a measure of symptom severity, with higher scores (range: 0-60) indicating greater depressive symptoms.
Change in anxiety and worry | At the baseline survey (1 day before the intervention begins), at the post-intervention survey (2 days after the final writing assignment), and and at the 2-week follow-up
  Symptoms of anxiety over the past week will be measured at baseline, post-intervention, and the 2-week follow-up via the 7-item Generalized Anxiety Disorder- 7 (GAD-7). Higher scores on the GAD-7 (range: 0-21) indicate greater severity of symptoms. Three additional items were added by the investigators to assess worry about vocational future: "I worry that I won't finish my degree," "I worry about what I will do after I finish my degree," and "I worry that I am not prepared for what comes after college (e.g., getting a job, graduate school)." These items are scored on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree), with higher scores indicating greater worry (range: 3-15).
Change in loneliness | At the baseline survey (1 day before the intervention begins), at the post-intervention survey (2 days after the final writing assignment), and and at the 2-week follow-up
  Feelings of loneliness over the past week will be measured at baseline, post-intervention, and the 2-week follow-up via the 8-item UCLA Loneliness Scale- Short Form 8. A higher overall score (range: 8-32) indicates greater feelings of loneliness.
Change in physical symptoms and health-care center visits | At the baseline survey (1 day before the intervention begins), at the post-intervention survey (2 days after the final writing assignment), and and at the 2-week follow-up
  Frequency of experiencing common physical symptoms (e.g., runny nose) over the past week will be measured at baseline, post-intervention, and the 2-week follow-up via a 13-item adapted version of the Pennebaker Inventory of Limbic Languidness (PILL). This measure includes 10-items assessing physical symptoms (range: 0-70), such as headache, shortness of breath, and coughing/sore throat, and 3-items assessing overall feelings of sickness ("how many days have you been sick?") and healthcare utilization ("how many visits have you made to the student health center?"). Greater scores indicate more physical symptoms/feelings of illness.
Change in sleep disturbance | At the baseline survey (1 day before the intervention begins), at the post-intervention survey (2 days after the final writing assignment), and and at the 2-week follow-up
  Sleep disturbance over the past week will be measured using the 4-item PROMIS Sleep Disturbance Scale at baseline, post-intervention, and the 2-week follow-up. Scores range from 4 to 20, with higher scores indicating more disturbance.
Change in social support | At the baseline survey (1 day before the intervention begins), at the post-intervention survey (2 days after the final writing assignment), and and at the 2-week follow-up
  Social support will be measured at baseline, post-intervention, and the 2-week follow-up using the 21-item 2-way Social Support Scale. This scale measures 4 dimensions of social support: instrumental support received, instrumental support given, emotional support received, and emotional support given. A higher total score (range: 0-105) indicates more feelings of perceived support.
Change in generativity | At the baseline survey (1 day before the intervention begins), at the post-intervention survey (2 days after the final writing assignment), and and at the 2-week follow-up
  Feelings of generativity will be measured at baseline, post-intervention, and the 2-week follow-up using the 13-item Generativity Scale. This measure consists of two subscales: generative desire and generative achievement, with higher scores (range: 13-78) indicating greater desire/achievement.
Change in positive and negative affect | At the baseline survey (1 day before the intervention begins), at the post-intervention survey (2 days after the final writing assignment), and and at the 2-week follow-up
  Daily reports of positive and negative affect will be assessed at baseline, post-intervention, the 2-week follow-up, and at each writing session using the 10-item positive affect subscale and 10-item negative affect subscales of the Positive and Negative Affect Schedule (PANAS-X). Two additional adjectives were also included, happy and calm. Greater scores indicate higher feelings of positive (range: 10-50) and negative affect (range: 10-50).
Change in fulfillment of psychological needs | At the baseline survey (1 day before the intervention begins), at the post-intervention survey (2 days after the final writing assignment), and and at the 2-week follow-up
  Fulfillment of psychological needs will be measured at baseline, post-intervention, the 2-week follow-up, and at each writing session using the 9-item Balanced Measure of Psychological Needs. This item has three subscales: autonomy, connectedness, and relatedness, with higher scores (range: 9-45) indicating greater needs satisfaction.

OTHER OUTCOMES:
Prosocial Tendencies (Moderator) | At the baseline survey (1 day before the intervention begins)
  Frequency of engaging in prosocial acts will be measured at baseline using the 20-item Self-Report Altruism Scale. Higher scores (range: 20-100) indicate more engagement in prosocial acts (e.g., helping a classmate with an assignment).

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No